CLINICAL TRIAL: NCT00005198
Title: Survival After Myocardial Infarction in A Biethnic Texas Community (Corpus Christi Heart Project)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1077; R01HL038429 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2001-08

CONDITIONS: Cardiovascular Diseases; Hypertension; Coronary Disease; Myocardial Infarction
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Coronary Disease; Myocardial Infarction

SUMMARY:
To determine the natural history of coronary heart disease in the biethnic community of Corpus Christi, Texas.

DETAILED DESCRIPTION:
BACKGROUND:

The decline in coronary heart disease mortality in the United States may be due to decreasing incidence of clinically apparent coronary heart disease or increasing survival from its first clinical appearance or both. Prior to 1987, few data were available to confirm either one directly. However, increased risk, decreased medical care, or both may predispose the Mexican-American population to increased recurrence of myocardial infarction and decreased post myocardial infarction survival, and an overall greater mortality among survivors of myocardial infarction, than are observed for Anglos in the same community setting. The significance of the potential results lies most importantly in the following aspects of this research: estimation of the community-based incidence of hospitalization for suspect, definite or possible myocardial infarction; precise determination of recurrence rates and survival curves after myocardial infarction in community-wide hospital-based cohorts; analysis of the relation of the above to risk status as ascertained at hospitalization and to health care and preventive practices assessed periodically post-myocardial infarction; and comparison of these observations between Anglos and Mexican-Americans, a group of special interest and concern because of expected differences in natural history of coronary heart disease and near total lack of the relevant data.

DESIGN NARRATIVE:

Patients hospitalized for acute coronary heart disease (CHD) in seven acute care hospitals in Nueces County, Texas were identified by active concurrent case registration. Baseline data on clinical, prognostic and sociodemographic characteristics of these patients at the time of the event were collected from the medical record and by interview with the patient. Patients with events meeting diagnostic criteria for acute myocardial infarction (MI) were followed directly through contacts at three months post-discharge and at the anniversary of discharge thereafter to ascertain vital status and to collect information about recurrent myocardial infarction, other changes in health status, and health care practices in the interim. Endpoints included all-cause mortality and deaths attributed to coronary heart disease, and fatal and non-fatal myocardial infarction. Data analysis included examination of survival and recurrence of myocardial infarction for the entire cohort of myocardial infarction patients and within ethnic groups; evaluation of potential prognostic factors within and between ethnic groups; and comparison of survival and myocardial infarction recurrence between ethnic groups after adjustment for both baseline and time-dependent covariates.

The study was renewed in 1992 to continue to identify hospitalized MI and CHD mortality as well as angioplasty, and bypass surgery among Mexican-Americans and non-Hispanic Whites. The investigators calculated incidence rates for hospitalized MI, for the use of cardiac revascularization, and rates for post-MI mortality, and for both all cause and CHD mortality in the community. They also described trends in these aspects of CHD over an eight year period and determined if ethnic differences existed.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1987-04; Study Completion 1998-03 (Actual)

REFERENCES:
- [Background] Goff DC Jr, Varas C, Ramsey DJ, Wear ML, Labarthe DR, Nichaman MZ. Mortality after hospitalization for myocardial infarction among Mexican Americans and non-Hispanic whites: the Corpus Christi Heart Project. Ethn Dis. 1993 Winter;3(1):55-63. PMID 8508105
- [Background] Orlander PR, Goff DC, Morrissey M, Ramsey DJ, Wear ML, Labarthe DR, Nichaman MZ. The relation of diabetes to the severity of acute myocardial infarction and post-myocardial infarction survival in Mexican-Americans and non-Hispanic whites. The Corpus Christi Heart Project. Diabetes. 1994 Jul;43(7):897-902. doi: 10.2337/diab.43.7.897. PMID 8013754
- [Background] Nichaman MZ, Wear ML, Goff DC Jr, Labarthe DR. Hospitalization rates for myocardial infarction among Mexican-Americans and non-Hispanic whites. The Corpus Christi Heart Project. Ann Epidemiol. 1993 Jan;3(1):42-8. doi: 10.1016/1047-2797(93)90008-r. PMID 8287155
- [Background] Goff DC Jr, Nichaman MZ, Ramsey DJ, Meyer PS, Labarthe DR. A population-based assessment of the use and effectiveness of thrombolytic therapy. The Corpus Christi Heart Project. Ann Epidemiol. 1995 May;5(3):171-8. doi: 10.1016/1047-2797(94)00103-z. PMID 7606305
- [Background] Blumberg MS. Re: "Greater case-fatality after myocardial infarction among Mexican Americans and women than among non-Hispanic whites and men: The Corpus Christi Heart Project". Am J Epidemiol. 1995 Mar 1;141(5):478-80. doi: 10.1093/oxfordjournals.aje.a117453. No abstract available. PMID 7794339
- [Background] Labarthe DR: Changing Patterns in the Epidemiology of Coronary Artery Disease: Trends in Survival After Myocardial Infarction. In: Long-Term Management of Patients After Myocardial Infarction. Kappagoda CT, Greenwood PV, (Eds), Pages 17-30, 1987
- [Background] Annegers JF, Hauser WA, Shirts SB, Kurland LT. Factors prognostic of unprovoked seizures after febrile convulsions. N Engl J Med. 1987 Feb 26;316(9):493-8. doi: 10.1056/NEJM198702263160901. PMID 3807992
- [Background] Slater CH, Green LW, Vernon SW, Keith VM. Problems in estimating the prevalence of physical activity from national surveys. Prev Med. 1987 Jan;16(1):107-18. doi: 10.1016/0091-7435(87)90010-7. PMID 3823009
- [Background] Slater CH, Carlton B, Ramirez G, Ashton C: Heart Disease, Strategies for Prevention. Eval Health Prof, 10(3):255-286, 1987
- [Background] Goff DC Jr, Ramsey DJ, Labarthe DR, Nichaman MZ. Greater case-fatality after myocardial infarction among Mexican Americans and women than among non-Hispanic whites and men. The Corpus Christi Heart Project. Am J Epidemiol. 1994 Mar 1;139(5):474-83. doi: 10.1093/oxfordjournals.aje.a117030. PMID 8154471
- [Background] Goff DC Jr, Ramsey DJ, Labarthe DR, Nichaman MZ. Acute myocardial infarction and coronary heart disease mortality among Mexican Americans and non-Hispanic whites in Texas, 1980 through 1989. Ethn Dis. 1993 Winter;3(1):64-9. PMID 8508106
- [Background] Goff DC, Nichaman MZ, Chan W, Ramsey DJ, Labarthe DR, Ortiz C. Greater incidence of hospitalized myocardial infarction among Mexican Americans than non-Hispanic whites. The Corpus Christi Heart Project, 1988-1992. Circulation. 1997 Mar 18;95(6):1433-40. doi: 10.1161/01.cir.95.6.1433. PMID 9118510
- [Background] Herholz H, Goff DC, Ramsey DJ, Chan FA, Ortiz C, Labarthe DR, Nichaman MZ. Women and Mexican Americans receive fewer cardiovascular drugs following myocardial infarction than men and non-Hispanic whites: the Corpus Christi Heart Project, 1988-1990. J Clin Epidemiol. 1996 Mar;49(3):279-87. doi: 10.1016/0895-4356(95)00572-2. PMID 8676174
- [Background] Farmer IP, Meyer PS, Ramsey DJ, Goff DC, Wear ML, Labarthe DR, Nichaman MZ. Higher levels of social support predict greater survival following acute myocardial infarction: the Corpus Christi Heart Project. Behav Med. 1996 Summer;22(2):59-66. doi: 10.1080/08964289.1996.9933765. PMID 8879457
- [Background] Goff DC Jr, Pandey DK, Chan FA, Ortiz C, Nichaman MZ. Congestive heart failure in the United States: is there more than meets the I(CD code)? The Corpus Christi Heart Project. Arch Intern Med. 2000 Jan 24;160(2):197-202. doi: 10.1001/archinte.160.2.197. PMID 10647758
- [Background] Morgenstern LB, Pandey DK, Smith MA, Ramsey D, Labarthe DR, Nichaman MZ. Greater stroke rate during hospitalization for acute heart disease among Mexican Americans than non-Hispanic whites. Neuroepidemiology. 1999;18(5):241-7. doi: 10.1159/000026218. PMID 10461049
- [Background] Meshack AF, Goff DC, Chan W, Ramsey D, Linares A, Reyna R, Pandey D. Comparison of reported symptoms of acute myocardial infarction in Mexican Americans versus non-Hispanic whites (the Corpus Christi Heart Project). Am J Cardiol. 1998 Dec 1;82(11):1329-32. doi: 10.1016/s0002-9149(98)00636-5. PMID 9856914
- [Background] Ramsey DJ, Goff DC, Wear ML, Labarthe DR, Nichaman MZ. Sex and ethnic differences in use of myocardial revascularization procedures in Mexican Americans and non-Hispanic whites: the Corpus Christi Heart Project. J Clin Epidemiol. 1997 May;50(5):603-9. doi: 10.1016/s0895-4356(97)80002-9. PMID 9180653
- [Background] Pladevall M, Goff DC, Nichaman MZ, Chan F, Ramsey D, Ortiz C, Labarthe DR. An assessment of the validity of ICD Code 410 to identify hospital admissions for myocardial infarction: The Corpus Christi Heart Project. Int J Epidemiol. 1996 Oct;25(5):948-52. doi: 10.1093/ije/25.5.948. PMID 8921479
- [Background] Steffen-Batey L, Nichaman MZ, Goff DC Jr, Frankowski RF, Hanis CL, Ramsey DJ, Labarthe DR. Change in level of physical activity and risk of all-cause mortality or reinfarction: The Corpus Christi Heart Project. Circulation. 2000 Oct 31;102(18):2204-9. doi: 10.1161/01.cir.102.18.2204. PMID 11056093
- [Background] Stimson WH, Blackstock JC. Synthesis of a pregnancy-associated alpha-macroglobulin by human leucocytes. Experientia. 1975 Mar 15;31(3):371-3. doi: 10.1007/BF01922593. No abstract available. PMID 1116554